CLINICAL TRIAL: NCT01321359
Title: A Randomized, Double-Blind, Parallel-Group, Vehicle-Controlled, Multicenter Study of NB-001 in the Treatment of Recurrent Herpes Labialis
Brief Title: A Multicenter Study of NB-001 in the Treatment of Recurrent Herpes Labialis
Acronym: SHaRCS
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: NanoBio Corporation (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: NB-001-004
Record Dates: First submitted 2011-03-22; First posted 2011-03-23 (Estimated); Last update posted 2013-05-23 (Estimated); Status verified 2013-05

CONDITIONS: Recurrent Herpes Simplex Labialis
MeSH Terms: conditions — Herpes Labialis

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Vehicle (Placebo Comparator): Vehicle
  Interventions: Drug: Vehicle versus NB-001
- Active (Active Comparator): Active NB-001(0.3%)
  Interventions: Drug: Vehicle versus NB-001

INTERVENTIONS:
Drug: Vehicle versus NB-001 — Topical, 5 times daily until investigator assessment of healing or a maximum of 4 days

SUMMARY:
Demonstrate the safety and efficacy of NB-001 in subjects with recurrent herpes labialis (RHL).

DETAILED DESCRIPTION:
This is a randomized, double-blind, two arm, parallel-group, vehicle-controlled, multi-center study of NB-001. The study is designed to demonstrate the safety and efficacy of NB-001 in subjects with RHL. Approximately 850 subjects who meet all eligibility criteria will be randomized in the study. Subjects will begin treatment as soon as they experience the onset of cold sore symptoms. Treatment will be applied 5 times daily, approximately 3-4 hours apart while awake. Treatment will continue until the investigator assesses the primary lesion complex as healed or a maximum of 4 days.

Clinic visits will occur on a daily basis until the investigator determines that the primary lesion complex has healed or a maximum of 15 clinic visits. At daily clinic visits, the investigator will make efficacy assessments of the primary lesion complex; safety and tolerability assessments of NB-001 following topical administration will also be assessed daily. Subjects will make daily assessments of therapy.

At the End of Study, the investigator will make a global assessment of therapy. The subject will make global assessments of therapy and social impact.

ELIGIBILITY:
Inclusion Criteria:

* A Healthy man or woman 18 years of age or older. Women who are pregnant, lactating or may become pregnant may (at the investigator's discretion) be included in the study.
* Have recurrent herpes labialis as defined by a history of three (3) or more cold sore recurrences on the lips and/or skin surrounding the lips in the previous 12 months;
* Have the majority of their cold sore recurrences proceeded by a well defined history of prodromal symptoms.

Exclusion Criteria:

* Subjects with severe chronic illness
* Received (within the last 6 months) or receiving chemotherapy;
* Significant skin disease on the face
* Previously received herpes vaccine;
* Active alcohol or drug abuse;
* Prior randomization into any NanoBio study;
* Known allergies to topical creams, ointments or other topical medications.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 907 (Actual)
Dates: Start 2011-04; Primary Completion 2012-01 (Actual); Study Completion 2012-01 (Actual)

PRIMARY OUTCOMES:
Time of Healing of the primary lesion complex | Days
  Time to healing of the primary lesion complex (in days or fraction thereof) as assessed by the investigator. Time to healing is the time from application of the first dose to investigator assessed healing

SECONDARY OUTCOMES:
Proportion of subjects in whom the primary lesion complex does not progress beyond the Papule/Edema Stage. | First Post-Treatment Visit
  Proportion of subjects in whom the primary lesion complex does not progress beyond the Papule/Edema Stage. This analysis will be performed in the cohort of subjects whose primary lesion complex is assessed as being in the Prodrome (pain, burning, tingling, itching, redness, swelling, or a tight sensation of the lip), Erythema/Macule, Papule/Edema, or Aborted Stage by the investigator at the first post-treatment visit.

CONTACTS AND LOCATIONS:
Locations (35):
- United States (35):
  - Radiant Research, Inc, Chandler, Arizona
  - Radiant Research, Inc, Scottsdale, Arizona
  - ACR-Phase 1, LLC., Anaheim, California
  - Northern California Research, Sacramento, California
  - Medical Center for Clinical Research, San Diego, California
  - Radiant Research, Inc, Santa Rosa, California
  - Westlake Medical Research, Westlake Village, California
  - Longmont Medical Research Network, Longmont, Colorado
  - Avail Clinical Research, LLC, DeLand, Florida
  - Clinical Study Center, Fort Myers, Florida
  - AGA Clinical Trials, Hialeah, Florida
  - Orlando Clinical Research Center, Orlando, Florida
  - Progressive Medical Research, Port Orange, Florida
  - Radiant Research, Inc, Atlanta, Georgia
  - Advanced Clinical Research, Meridan, Idaho
  - MediSphere Medical Research Center, LLC, Evansville, Indiana
  - Radiant Research, Inc., Overland Park, Kansas
  - Central Kentucky Research Associates, Inc., Lexington, Kentucky
  - Michigan Center for Research Corp, DBA Michigan Center for Skin Care Research, Clinton Township, Michigan
  - Radiant Research, Inc., Edina, Minnesota
  - Pioneer Clinical Research, LLC, Bellevue, Nebraska
  - Regional Clinical Research, Inc., Endwell, New York
  - Physicians' Research, Inc., Zanesville, Ohio
  - Westover Heights Clinic, Portland, Oregon
  - Paddington Testing Co, Inc, Philadelphia, Pennsylvania
  - Primary Physicians Research, Pittsburgh, Pennsylvania
  - Radiant Research, Inc, Greer, South Carolina
  - Coastal Carolina Research Center, Mt. Pleasant, South Carolina
  - Clinical Research Associates, Inc., Nashville, Tennessee
  - J&S Studies, Inc., College Station, Texas
  - Radiant Research-Dallas North, Dallas, Texas
  - Benchmark Research, Fort Worth, Texas
  - Research Across America, Plano, Texas
  - Intermountain Clinical Research, Draper, Utah
  - New River Valley Research Institute, Christiansburg, Virginia